CLINICAL TRIAL: NCT02774070
Title: Characteristics of Rheumatoid Arthritis Patients With Asymptomatic Versus Symptomatic Atlantoaxial Joint Affection Detected by Plain X-ray and Magnetic Resonance Imaging
Brief Title: Characteristics of Rheumatoid Arthritis Patients With Atlantoaxial Synovitis Detected by Plain X-ray and MRI
Acronym: MRI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial support
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nisreen Adel Abbas, Doctor of diagnostic radiology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Rheumatoid AAJ
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Neck Pain
Keywords: AAJ RA MRI synovitis
MeSH Terms: conditions — Neck Pain | interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symptomatic atlantoaxial joint affection (Other): Undergo plain X-ray and magnetic resonance imaging
  Interventions: Radiation: Plain X-ray; Radiation: Magnetic resonance imaging
- Asymptomatic atlantoaxial joint aff. (Other): Undergo plain X-ray and magnetic resonance imaging
  Interventions: Radiation: Plain X-ray; Radiation: Magnetic resonance imaging

INTERVENTIONS:
Radiation: Plain X-ray — antero-posterior, lateral neutral, flexion, extension and open-mouth views
Radiation: Magnetic resonance imaging — Magnetic resonance imaging sagittal T1W,T2W and STIR, axial T1W and coronal T2W and post contrast sagittal and axial sequences

SUMMARY:
This study detects the presence of atlantoaxial joint affection in symptomatic versus asymptomatic rheumatoid arthritis patients revealed by plain X-ray and magnetic resonance imaging of the cervical spine

DETAILED DESCRIPTION:
Atlantoaxial joint affection in rheumatoid arthritis patients may have life-threatening complications if not detected early. It may not be detected unless it becomes symptomatic. However, asymptomatic atlantoaxial joint affection is not uncommon. Investigators will try to detect atlantoaxial joint affection at an early stage and its relation to symptomatology and other disease criteria. So investigators will use conventional plain X-ray examination combined with magnetic resonance imaging of the cervical spine to detect soft tissue as well as bony changes of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients complaining or not complaining of atlantoaxial affection symptomatology

Exclusion Criteria:

* Pregnant females
* Patients with pacemakers or metallic bony plates.
* Patients that have claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Prevelance of atlantoaxial joint affection in clinically and laboratory proven rheumatoid arthritis patients | 3 months
  Prevelance of atlantoaxial joint affection in symptomatic versus asymptomatic rheumatoid arthritis patients

CONTACTS AND LOCATIONS:
Overall Officials: Nisreen A Abbas, Doctor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yurube T, Sumi M, Nishida K, Miyamoto H, Kohyama K, Matsubara T, Miura Y, Hirata H, Sugiyama D, Doita M. Accelerated development of cervical spine instabilities in rheumatoid arthritis: a prospective minimum 5-year cohort study. PLoS One. 2014 Feb 18;9(2):e88970. doi: 10.1371/journal.pone.0088970. eCollection 2014. PMID 24558457
- [Background] Nazarinia M, Jalli R, Kamali Sarvestani E, Farahangiz S, Ataollahi M. Asymptomatic atlantoaxial subluxation in rheumatoid arthritis. Acta Med Iran. 2014;52(6):462-6. PMID 25130155